CLINICAL TRIAL: NCT04181229
Title: Deep Brain Stimulation After Failed Vagal Nerve Stimulation for the Treatment of Drug-Resistant Epilepsy in Children
Brief Title: Deep Brain Stimulation Post Failed Vagal Nerve Stimulation
Acronym: DBSpostVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, George Ibrahim, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB1000063803
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy, Drug Resistant
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Treatment arm - DBS Control arm - Continued VNS (optimization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBS Treatment (Experimental): Patients in the treatment arm will receive DBS of bilateral centromedian nucleus (2 electrodes per patient). DBS is a standard of care treatment option for drug-resistant epilepsy patients who have previously failed VNS at 12 months or more after instigation and optimization of therapy.
  Interventions: Procedure: Deep brain stimulation
- Continued VNS (control) (No Intervention): For the control arm, the patients will be monitored for one year with the same standard assessments used for the measurement of seizure frequency and severity. No changes will be made to these patients' treatment plan. These patients will be placed on a wait list for CM-DBS treatment of seizures if that is the desire of the patient and/or their family. After the 12 months of observation, these patients can choose to undergo DBS surgery.

INTERVENTIONS:
Procedure: Deep brain stimulation — Patients will receive surgical implantation of the Medtronic DBS device (Device # 37601). Two (2) electrodes will be implanted bilaterally in the centromedian nucleus.
  Arms: DBS Treatment

SUMMARY:
This is a multicenter, non-blinded, patient preference comparative trial for efficacy of deep brain stimulation (DBS) on drug-resistant epilepsy compared to continued vagal nerve stimulation (VNS) optimization in children with failed VNS. The two conditions being compared are therefore DBS (treatment) versus VNS (control). Fifty (50) patients will be recruited and enrolled in this pilot study (25 from The Hospital for Sick Children and 50 from CHU Sainte-Justine).

DETAILED DESCRIPTION:
For children with epilepsy that have failed pharmacological and alternative treatments (drug-resistant epilepsy; [DRE]), surgical interventions may be considered. This includes vagus nerve stimulation (VNS) and deep brain stimulation (DBS). VNS for the treatment of DRE in children is an established and widely used treatment. Unfortunately, the positive response to VNS rate (>50% reduction in seizures) is not consistent, ranging from 26-55% in pediatric epilepsy patients. In children with failed VNS, defined as no improvement in seizure control after at least 1 year of treatment, they may undergo DBS as a recommended therapy. DBS is a safe and established treatment for various childhood neurological conditions and the indications for DBS in children continue to expand. It is currently unknown which children may benefit from DBS after failed VNS.

As a patient-preference randomized trial, patients and their parents will be introduced to the options of continuing with current VNS management (control arm) or trialing DBS (treatment arm). Patients and their parents will fall into three possible groups according to preference and willingness for randomization.

i) Patients with no strong preferences and consent to randomization ii) Patients with a preference, yet still consent to randomization iii) Patients who refuse randomization and opt for enrollment in a specific arm

Patients in the treatment arm will receive DBS of the centromedian nucleus. The centromedian nucleus is believed to reduce electrocortical activity in generalized epilepsy. The investigators hypothesize that stimulating this target will lead to a decrease in seizure severity and frequency in patients who have failed VNS; in comparison with patients who will have continued VNS treatment and optimization. Patients in the control arm will continue to be observed for 12 months with no change to their treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients 8 years of age and over but not including 18 year olds.
2. Diagnosis of drug-resistant epilepsy with failure after trial of two anti-epileptic medications (as defined by Kwan et al. 20093). All children screened for entry into the study will be re-diagnosed by a neurologist prior to entry.
3. Failure of vagal nerve stimulation, defined as the same or increased frequency and severity of seizures at 12 months or more after instigation and optimization of therapy. Failure is defined objectively and subjectively. Objective evidence includes caregiver logs, clinician assessment, or neuromonitoring if the clinician has documented a baseline status prior to instigation of vagal nerve stimulation. Subjective measures include family or patient opinion that seizure frequency or severity has not improved.
4. Parents or legal guardians, including caregivers, who are informed and able to give written consent.
5. Ability to comply with all testing, follow-ups and study appointments and protocols for 12 months following the end of the duration of the study.

Exclusion Criteria:

1. Substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
2. Any contraindication to MRI scanning. A preoperative MRI scan is essential to planning DBS and therefore any contraindication to MRI is a contraindication to enrollment in the study.
3. Unwillingness or inability to return to SickKids for follow-up visits.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Seizure reduction after DBS surgery | Assessed post surgery up to 1 year
  Measured by the Class on the Engel Epilepsy Surgery Outcome Scale, where:
  Class I: Free of disabling seizures IA: Completely seizure-free since surgery IB: Non disabling simple partial seizures only since surgery IC: Some disabling seizures after surgery, but free of disabline seizures for at least 2 years ID: Generalized convulsions with antiepileptic drug withdrawal only Class II: Rare disabling seizures ("almost seizure-free") IIA: Initially free of disabling seizures but has rare seizures now IIB: Rare disabling seizures since surgery IIC: More than rare disabling seiuzres after surgery, but rare seizures for at least 2 years IID: Nocturnal seizures only Class III: Worthwhile improvement IIIA: Worthwhile seiuzre reduction IIIB: Prolonged seiuzre-free intervals amounting to greater than half the follow-up period, but not less than 2 years Class IV: No worthwhile improvement IVA: Significant seizure reduction IVB: No appreciable change IVC: Seizures worse
Seizure reduction after VNS surgery | Assessed post surgery up to 1 year
  Measured by the Class on the McHugh Scale, where:
  Class I (80-100% reduction in seizure frequency) Class II (50-79% reduction in seizure frequency) Class III (< 50% reduction in seizure frequency) Class IV (Magnet benefit only) Class V (No improvement)

SECONDARY OUTCOMES:
Change in patient-perceived seizure severity | Assessed pre surgery and post surgery up to 1 year
  Measured by the Liverpool Seizure Severity Scale (LSSS) which measures patients' own perceptions of changes in seizure severity. The LSSS is rated on a 4-point likert scale, where 1 represents "always" (worse outcome) and 4 represents "never" (better outcome).
Change in parent-perceived seizure severity | Assessed pre surgery and post surgery up to 1 year
  Measured by the Hague Seizure Severity (HASS) scale which measures parents' perceptions of changes in seizure severity. The HASS is measured on a 4 point likert-scale, where 1 represents "always" (worse outcome) and 4 represents "never" (better outcome).
Change in self-reported quality of life | Assessed pre surgery and post surgery up to 1 year
  Measured by the Quality of Life in Epilepsy for Adolescents scale (QOLIE-AD-48), a two-part scale. Part 1 measures general health on a 5 point scale where 1 represents "excellent" (better outcome) and 5 represents "poor" (worse outcome). Part 2 measures effects of epilepsy and antiepilepsy medications on a 5 point scale where 1 represents "very often" (worse outcome) and 5 represents "never" (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: George Ibrahim, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.